CLINICAL TRIAL: NCT01713088
Title: A Trial of Multisystemic Therapy in UK a Statutory Therapeutic Intervention for Young Offenders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Brandon Centre, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MSTBC2012; MSTBC2012 (Other: Brandon Centre)
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Participants Are Male and Female Adolescents 13-16 Years at Risk for Continuing to Commit Criminal Offences.
Keywords: multisystemic therapy, RCT, young offenders, U.K.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multisystemic therapy (Experimental): MST is a family- and community-based intervention that establishes close contact with families to understand and deal with the factors that cause the young person's antisocial behaviour. The intervention targets the individual's adjustment, family relationships, school functioning and peer group affiliations. Therapists help caretakers develop skills to intervene and operate changes in important domains such as young person's individual adjustment, their family relationships, school functioning, and peer group affiliations.
  Interventions: Other: Multisystemic therapy
- YOT (usual services) (Active Comparator): YOT intervention consisted of services currently available to young offenders in accordance with the Youth Justice Board National Standards.These services included supporting the young person to re-engage with education, with substance misuse problems and anger management; training them in social problem-solving skills; and programs to decrease vehicle-crime, violent-offending and knife crime. The treatments were delivered by professional social workers, specialist therapists or probation officers.
  Interventions: Other: YOT (usual services)

INTERVENTIONS:
Other: Multisystemic therapy
  Arms: Multisystemic therapy
Other: YOT (usual services)
  Arms: YOT (usual services)

SUMMARY:
To evaluate whether Multisystemic Therapy (MST) is more effective in reducing youth offending and out-of-home placement in a large, ethnically diverse, urban U.K. sample than an equally comprehensive management protocol; to determine whether MST leads to broader improvements in youth sociality and in mediators believed to be responsible for change in MST.

ELIGIBILITY:
Inclusion Criteria:

* age between 13 and 16 years;
* living in the home of and being brought up by a parent or principal caretaker;
* on a court referral order for treatment or a supervision order of at least 3 months' duration, or, following imprisonment, on license in the community for at least 6 months.

Exclusion Criteria:

* being a sex offender;
* presented only with substance misuse;
* diagnosed with a psychotic illness or posed a risk to trial personnel;
* incompatible agency involvement (e.g., ongoing care proceedings).

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2003-11; Primary Completion 2010-09 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Change in offending behavior based on police records of criminal offenses committed | baseline and 6, 12, 18, 24, 30 and 36 months post randomization
  The number of records of offending behavior (count data) was obtained, and 6-month periods free of any offending behavior were also recorded (binary data). Records were obtained from the National Young Offender Information System (YOIS) database. YOIS records detail offence information, court appearances, criminal orders, police custody records, and arrest rates.

SECONDARY OUTCOMES:
self- and parent-rated symptoms of antisocial behavior, delinquency-linked cognitions, personality functioning, and parenting variables | baseline and 6 months after randomization
  Antisocial behavior was assessed using the Self-Report of Youth Behavior (SRYB), a brief, valid measure of the prevalence and incidence in pre-adolescent and adolescent children of delinquent behavior such as vandalism, theft, burglary, and fraud; and the delinquency and aggression subscales of the Youth Self-Report (YSR) and the parent-completed Child Behavior Checklist (CBCL).

OTHER OUTCOMES:
Antisocial Beliefs and Attitudes Scale (ABAS) | Baseline and 6 months after randomization
Antisocial Process Screening Device (APSD) | Baseline and 6 months after randomization
Measure of youth's involvement with delinquent peers (IDP) | Baseline and 6 months after randomization
Measure of Positive Parenting and Disciplinary Practices, Parent Monitoring and Supervision | Baseline and 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The Brandon Centre, London, London, United Kingdom

REFERENCES:
- [Result] Butler S, Baruch G, Hickey N, Fonagy P. A randomized controlled trial of multisystemic therapy and a statutory therapeutic intervention for young offenders. J Am Acad Child Adolesc Psychiatry. 2011 Dec;50(12):1220-35.e2. doi: 10.1016/j.jaac.2011.09.017. Epub 2011 Nov 6. PMID 22115143
- See also: Related Info — http://www.brandon-centre.org.uk/